CLINICAL TRIAL: NCT06079151
Title: Physiological Evaluation of the Hemodynamic Effects of Nasal High Flow in Patients Being Explored by Right Heart Catheterisation and Echocardiography for Suspected or Followed Precapillary Pulmonary Hypertension
Brief Title: Hemodynamic Effect of Nasal High-flow in Patients Suspected or Followed for a Precapillary Pulmonary Hypertension
Acronym: HighFlowHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ADIR Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HighFlowHD
Record Dates: First submitted 2023-08-22; First posted 2023-10-12 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Pulmonary Hypertension
Keywords: High-flow nasal cannula therapy; Hemodynamic monitoring; Echocardiography; right heart catheterization
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: All patients will be randomly allocated into two groups using the block randomization technique (4 or 8 according to an equiprobable distribution) in a 1:1 ratio. The randomisation will be performed at the begining of the catheterization procedure. In the first arm, the patient will successively receive 30 L/min then 50 L/min of room air. In the second arm, the patient will successively receive 50 L/min then 30 L/min of room air.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal high-flow 30 L/min and then 50 L/min (Experimental): The patient will be placed successively under nasal high-flow 30 L/min during 20 min and then 50 L/min during 20 min.
  Interventions: Device: Nasal high-flow
- Nasal high-flow 50 L/min and then 30 L/min (Experimental): The patient will be placed successively under nasal high-flow 50 L/min during 20 min and then 30 L/min during 20 min.
  Interventions: Device: Nasal high-flow

INTERVENTIONS:
Device: Nasal high-flow — Nasal high-flow is a respiratory technique which allows the administration of warmed and humidified air, associated with oxygen if necessary

SUMMARY:
In this study, the investigators aim to describe the hemodynamic consequences of nasal high-flow measured during right heart catheterization and echocardiography. The research hypothesis is that nasal high-flow would increase cardiac output in patients with pulmonary hypertension. The concomitant echocardiography will allow to describe its sensibility to detect cardiovascular consequences of nasal high-flow.

ELIGIBILITY:
Inclusion Criteria:

- patient addressed for right heart catheterization for pulmonary hypertension suspicion or follow-up.

Exclusion Criteria:

* necessity of FiO2 >21% during right heart catheterization
* intracardiac shunt
* grade 4 tricuspid insufficiency
* complete arrhythmia due to atrial fibrillation
* Pregnant or breastfeeding women or women of childbearing age without an effective method of contraception
* protected adult patient (tutorship or curatorship)
* patient deprived of liberty by court or administrative decision
* refusal of patient participation or consent
* patient for whom the measurement of pulmonary arterial pressures during right heart catheterization is impossible
* patient for whom, during the etiological assessment of pulmonary hypertension, the diagnosis of precapillary pulmonary hypertension cannot be confirmed and classified in groups 1, 3 or 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min

SECONDARY OUTCOMES:
cardiac output | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
cardiac output | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
Right atrial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
Right atrial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
Right atrial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
systolic pulmonary arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
systolic pulmonary arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
systolic pulmonary arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
diastolic pulmonary arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
diastolic pulmonary arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
diastolic pulmonary arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
mean pulmonary arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
mean pulmonary arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
mean pulmonary arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
capillary wedge pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
capillary wedge pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
capillary wedge pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
pulmonary vascular resistance | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
pulmonary vascular resistance | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
pulmonary vascular resistance | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
central venous oxygen saturation | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
central venous oxygen saturation | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
central venous oxygen saturation | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
heart rate | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
heart rate | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
heart rate | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
systolic arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
systolic arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
systolic arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
diastolic arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
diastolic arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
diastolic arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
mean arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
mean arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
mean arterial pressure | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
systolic ejection volume | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
systolic ejection volume | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
systolic ejection volume | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
respiratory rate | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
respiratory rate | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
respiratory rate | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
pulse oxygen saturation | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 50L/Min FiO2 21% as compared to room air
pulse oxygen saturation | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30L/Min FiO2 21% as compared to room air
pulse oxygen saturation | During the intervention, at isotime
  Changes measured during cardiac catheterization under nasal high-flow 30 and 50 L/min
Consequences of nasal high-flow 50 and 30 L/min FiO2 21% on echocardiographic parameters. | During the intervention, at isotime
  Cardiac output, inferior vena cava diameter and collapsibiliy, systolic pulmoanry arterial pressure, tricuspid regurgitation velocity,tricuspid annular plane systolic excursion, right ventricule strain, tricuspid S wave, right on left ventricular telediastolic surface ratio, left ventricular ejection fraction, mitral doppler, mitral S wave, respiratory variability of E mitral wave
systolic pulmonary arterial pressure measured by catheterization and echocardiography. | During the intervention, at isotime
  Concordance and correlation of hemodynamic parameters measured by catheterization and echocardiography.
capillary wedge pressure measured by catheterization and echocardiography. | During the intervention, at isotime
  Concordance and correlation of hemodynamic parameters measured by catheterization and echocardiography.
right atrial pressure measured by catheterization and echocardiography. | During the intervention, at isotime
  Concordance and correlation of hemodynamic parameters measured by catheterization and echocardiography.
cardiac output measured by catheterization and echocardiography. | During the intervention, at isotime
  Concordance and correlation of hemodynamic parameters measured by catheterization and echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Elise ARTAUD-MACARI, MD, Principal Investigator — ADIR Association
Locations (1):
- ROUEN university hospital, Rouen, France